CLINICAL TRIAL: NCT03231904
Title: The Correlation Between Gestational Age and Maternal and Fetal Levels of LIF and ACTH
Brief Title: Maternal and Fetal Adrenocorticotropic Hormone (ACTH) and Leukemia Inhibitory Factor (LIF) and Gestational Age
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Yuval Ginsberg, MD, Principal Investigator, Rambam Health Care Campus
Other Study IDs: 0508-16-RMB
Record Dates: First submitted 2017-07-01; First posted 2017-07-27 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Abortion, Legal
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fetal and maternal blood samples for ACTH and LIF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood test — blood samples will be taken for maternal and fetal levels of ACTH and LIF

SUMMARY:
In 2010, Simamura et al have demonstrated in a rat model that one of the pro-inflammatory cytokine belonging to the Interleukin-6 family cytokines, LIF, is required for the proliferation of neuronal progenitor cells in the cerebrum. They have shown that maternal LIF induces ACTH from the placenta, which in turn stimulates fetal nucleated red blood cells to secrete LIF, leading finally to neurogenesis in the fetus As demonstrated recently in a mouse model, maternal inflammation suppress the physiological maternal- fetal LIF-ACTH-LIF signal, result in reduction of ACTH production from placenta, which lead to a reduction in LIF concentration in fetal Cerebrospinal fluid (CSF) and impaired proliferation of the neural stem/ progenitor cells and poor development of the fetal brain.

In the current study, the investigators will take fetal and maternal blood samples of fetuses undergoing termination of pregnancy (TOP) . Maternal samples will be acquired with the routine blood samples before performance of TOP , fetal blood samples will be acquired from the umbilical vessel after the termination has been completed , the blood samples will be analyzed for levels of LIF and ACTH and checked according to termination pregnancy week, Patients electronic files will be checked for relevant demographic and obstetric information.

DETAILED DESCRIPTION:
Study protocol:

In the current study, the investigators will take fetal and maternal blood samples of fetuses undergoing termination of pregnancy (TOP) . Maternal samples will be acquired with the routine blood samples before performance of TOP , fetal blood samples will be acquired from the umbilical vessel after the termination has been completed , the blood samples will be analyzed for levels of LIF and ACTH and checked according to termination pregnancy week, Patients electronic files will be checked for relevant demographic and obstetric information.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women undergoing termination of pregnancy in various gestational weeks.
* Pregnant women undergoing spontaneous abortion.

Exclusion Criteria:

•Intrauterine fetal death.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women undergoing termination of pregnancy
Study Population: Pregnant women undergoing termination of pregnancy for different reasons
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-08-10 (Estimated); Primary Completion 2017-11-30 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Maternal LIF levels during pregnancy | up to 6 months
  Differences in levels of LIF according to gestational age
Maternal ACTH levels during pregnancy | up to 6 months
  Differences in levels of ACTH according to gestational age
Fetal LIF levels during pregnancy | up to 6 months
  Differences in levels of LIF according to gestational age
Fetal ACTH levels during pregnancy | up to 6 months
  Differences in levels of ACTH according to gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Ginsberg, MD, Principal Investigator — Rambam Health Care Campus

IPD SHARING:
Plan to Share IPD: No